CLINICAL TRIAL: NCT00326118
Title: Study to Demonstrate Non-inferiority of GSK Biologicals' Hib-MenC With Priorix™, Versus MenC-CRM197 Vaccine With Hiberix™ & Priorix™ in Toddlers Primed With Hib But Not MenC & to Evaluate Persistence up to 5 Years After Vaccination.
Brief Title: Study in Toddlers to Demonstrate Non-inferiority of GSK Biologicals' Hib-MenC & to Evaluate Persistence up to 5 Years.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106445; 106446 (Other: GSK); 106449 (Other: GSK); 106450 (Other: GSK); 106452 (Other: GSK); 106454 (Other: GSK)
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Results first posted 2009-10-23 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: Meningococcal serogroup C diseases; H.influenzae type b diseases
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines; Measles-Mumps-Rubella Vaccine; Hiberix

ARMS (2):
- Meningitec + Hiberix Group (Active Comparator): Subjects received a single dose of Meningitec™ vaccine co-administered with Hiberix™ and Priorix™ vaccines. The Meningitec vaccine was administered intramuscularly in the left deltoid region, the Hiberix vaccine was administered intramuscularly in the left thigh region and the Priorix vaccine was administered subcutaneously in the right upper arm.
  Interventions: Biological: Priorix™; Biological: Hiberix™; Biological: Meningitec™
- Menitorix Group (Experimental): Subjects received a single dose of Menitorix™ vaccine co-administered with Priorix™ vaccine. Menitorix vaccine was administered intramuscularly in the left deltoid region and the Priorix vaccine was administered subcutaneously in the right upper arm.
  Interventions: Biological: Haemophilus influenzae type b and meningococcal serogroup C (vaccine); Biological: Priorix™

INTERVENTIONS:
Biological: Haemophilus influenzae type b and meningococcal serogroup C (vaccine) — One intramuscular dose at 12-18 months of age
  Other Names: Hib-MenC; Menitorix™
  Arms: Menitorix Group
Biological: Priorix™ — One subcutaneous dose at 12-18 months of age
Biological: Hiberix™ — One intramuscular dose at 12-18 months of age.
  Arms: Meningitec + Hiberix Group
Biological: Meningitec™ — One intramuscular dose at 12-18 months of age
  Arms: Meningitec + Hiberix Group

SUMMARY:
The purpose of the primary phase of the study is to demonstrate the non-inferiority of a single dose of GSK Biologicals' Haemophilus influenzae type b and meningococcal C (Hib-MenC) conjugate vaccine when given in the second year of life to subjects primed in infancy with a Hib vaccine, but not with a meningococcal serogroup C vaccine, versus commercially available Hib and MenC vaccines.

In the extension phase, at Years 1, 2, 3, 4 & 5, one blood sample is taken at each year to follow the antibody persistence up to 5 years after vaccination. No additional vaccine is administered during the extension phase. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This multicenter study is open and has 2 treatment groups with Hiberix™ + a commercially available MenC vaccine as active controls. Priorix™ is given concomitantly in both groups. In the primary phase, two blood samples are taken from all subjects for immunogenicity analyses: before and one month after vaccination. In the extension phase, at Year 1, 2, 3, 4 & 5, one blood sample is taken at each year to follow the antibody persistence up to 5 years after vaccination. No additional vaccine is administered during the extension phase.

ELIGIBILITY:
Inclusion Criteria:

Primary phase:

* Subjects whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 18 months of age at the time of vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her parents'/guardians knowledge.
* Having completed primary vaccination with two doses of Haemophilus influenzae type b outer membrane protein (Hib-OMP) containing vaccine OR three doses of diphtheria, tetanus, acellular pertussis and Haemophilus influenzae type b (DTPa/Hib) containing vaccine at least 6 months before the study start.

Long-term persistence phase:

- Having participated in the vaccination study 106445

Exclusion Criteria:

For the primary vaccination phase:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) or planned administration of immuno-suppressants or other immune-modifying drugs within six months prior to vaccination.
* Planned administration/administration of a vaccine not foreseen by the protocol during the period starting from 30 days before vaccination and ending 30 days after vaccination.
* Administration of a meningococcal vaccine not foreseen by the study protocol during the period starting at birth and ending at first dose.
* Previous administration of a booster dose of Hib vaccine.
* Previous vaccination against measles, mumps, rubella.
* History of H. influenzae type b, meningococcal serogroup C and/or confirmed measles, mumps or rubella diseases.
* Known exposure to measles, mumps or rubella within 30 days prior to the start of the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of neurological disorders or more than one episode of febrile convulsion.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Additional exclusion criteria for the long-term persistence phase: to be checked each year.

* Previous administration of a booster dose of Hib, meningococcal serogroup C vaccines.
* History of H. influenzae type b, meningococcal serogroup C diseases.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 433 (Actual)
Dates: Start 2006-06-01; Primary Completion 2007-11-01 (Actual); Study Completion 2007-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Australia (7):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Booy R, Richmond P, Nolan T, McVernon J, Marshall H, Nissen M, Reynolds G, Ziegler JB, Heron L, Lambert S, Caubet M, Mesaros N, Boutriau D. Immediate and longer term immunogenicity of a single dose of the combined haemophilus influenzae type B-Neisseria meningitidis serogroup C-tetanus toxoid conjugate vaccine in primed toddlers 12 to 18 months of age. Pediatr Infect Dis J. 2011 Apr;30(4):340-2. doi: 10.1097/INF.0b013e31820013d2. PMID 21068692
- [Background] Booy R, Richmond P, Nolan T, McVernon J, Marshall H, Nissen M, Reynolds G, Ziegler JB, Stoney T, Heron L, Lambert S, Mesaros N, Peddiraju K, Miller JM. Three-year antibody persistence and safety after a single dose of combined haemophilus influenzae type b (Hib)-Neisseria meningitidis serogroup C-tetanus toxoid conjugate vaccine in Hib-primed toddlers. Pediatr Infect Dis J. 2013 Feb;32(2):169-74. doi: 10.1097/INF.0b013e3182787bff. PMID 23080288
- [Background] Booy R et al. Immunogenicity and safety of the Hib-MenC-TT conjugate vaccine in Hib-primed toddlers: 3 year follow-up. Abstract presented at the 7th World Congress for World Society for Pediatric Infectious Diseases (WSPID). Melbourne, Australia, 16-19 November 2011.
- [Background] Booy R et al. Immunogenicity and safety of the Hib-MenC-TT conjugate vaccine in Hib-primed toddlers: 4 year follow-up. Abstract presented at the Communicable Diseases Network Australia - Communicable Diseases Control Conference 2013, Canberra, Australia, 19-20 March 2013.
- [Background] Booy R et al. Prolonged immunogenicity and safety of the HibMenC-TT conjugate vaccine in Hib-Primed toddlers. Abstract presented at the PHAA Communicable Disease Conference. Canberra, Australia, 4-6 April 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 106445 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106445 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106445 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106445 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106445 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106445 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of subjects completed in the previous period does not necessarily correspond to the amount of subjects who came back for the follow-up. These subjects were considered lost-to-follow-up.
Period: Active Phase
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Started | 324 | 109
Completed | 320 | 108
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1
Period: Year 1 Follow-up
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Started | 295 | 100
Completed | 295 | 100
Not Completed | 0 | 0
Period: Year 2 Follow-up
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Started | 270 | 92
Completed | 270 | 92
Not Completed | 0 | 0
Period: Year 3 Follow-up
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Started | 256 | 89
Completed | 256 | 89
Not Completed | 0 | 0
Period: Year 4 Follow-up
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Started | 228 | 80
Completed | 228 | 80
Not Completed | 0 | 0
Period: Year 5 Follow up
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Started | 217 | 78
Completed | 217 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menitorix Group | Meningitec + Hiberix Group | Total
Number analyzed (Participants) | 324 | 109 | 433
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.5 (0.94) | 12.5 (0.75) | 12.5 (0.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 42 | 192
  Male | 174 | 67 | 241

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Greater Than or Equal to 0.15 Micrograms Per Milliliter (µg/mL)
Description: Anti-PRP antibody concentration greater than or equal to 0.15 µg/mL is indicative of short-term protection.
Time Frame: 1 month after vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity which included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component for the blood sample taken 1 month after vaccination.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 292 | 100
Subjects | 292 | 100

2. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers Greater Than or Equal to 1:8 Titer
Description: rSBA-MenC titers greater than or equal to 1:8 titer are indicative of seroprotection.
Time Frame: 1 month after vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 281 | 98
Subjects | 280 | 98

3. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers Above the Cut-off Values
Description: rSBA-MenC titers cut-off values assessed were greater than or equal to (≥) 1:8 (indicative of seroprotection) and ≥ 1:128 titers.
  Functional anti-meningococcal serogroup C activity (SBA-MenC) was determined by a serum bactericidal test using rabbit complement. For SBA testing at a GlaxoSmithKline (GSK) laboratory up to Year 3 after vaccination, titres were expressed as the reciprocal of the dilution resulting in 50% inhibition. For SBA testing at the Public Health England (PHE), formerly known as Health Protection Agency (HPA), at Year 4, titres were expressed as the reciprocal of the last dilution resulting in at least 50% inhibition.
Time Frame: Prior to, 1 month, 1 year, 2 years, 3 years and 4 years after vaccination
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity (prior to and 1 month after vaccination) and the ATP cohort for analysis of persistence for Year 1, 2, 3 and 4 (1, 2, 3 and 4 years after vaccination), on subjects with available data for at least one tested antigen at the considered time point.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 281 | 98
Subjects
  ≥ 1:8 [Prior to vaccination] (N=255, 83) | 37 | 7
  ≥ 1:8 [1 year after vaccination] (N=249, 89) | 216 | 68
  ≥ 1:8 [2 years after vaccination] (N= 235, 86) | 164 | 52
  ≥ 1:8 [3 years after vaccination] (N= 226, 77) | 145 | 41
  ≥ 1:8 [4 years after vaccination] (N= 208, 73) | 26 | 9
  ≥ 1:128 [Prior to vaccination] (N=255, 83) | 15 | 3
  ≥ 1:128 [1 month after vaccination] (N=281, 98) | 247 | 89
  ≥ 1:128 [1 year after vaccination] (N=249, 89) | 117 | 37
  ≥ 1:128 [2 years after vaccination] (N= 235, 86) | 76 | 26
  ≥ 1:128 [3 years after vaccination] (N= 226, 77) | 58 | 22
  ≥ 1:128 [4 years after vaccination] (N= 208, 73) | 7 | 4

4. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers Above the Cut-off Values
Description: rSBA-MenC titers cut-off values assessed were greater than or equal to (≥)1:8 (indicative of seroprotection) and 1:128 titers. For SBA testing at the PHE at Year 5, titres were expressed as the reciprocal of the last dilution resulting in at least 50% inhibition.
Time Frame: 5 years after vaccination
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of persistence for Year 5, on subjects with available data for at least one tested antigen at the considered time point.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 195 | 68
Subjects
  ≥ 1:8 [5 years after vaccination] | 37 | 17
  ≥ 1:128 [5 years after vaccination ] | 12 | 7

5. Secondary Outcome: Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers
Description: Titers are given as Geometric Mean Titers (GMTs). Functional anti-meningococcal serogroup C activity (SBA-MenC) was determined by a serum bactericidal test using rabbit complement. For SBA testing at a GlaxoSmithKline (GSK) laboratory up to Year 3 after vaccination, titres were expressed as the reciprocal of the dilution resulting in 50% inhibition. For SBA testing at the PHE at year 4 after vaccination, titres were expressed as the reciprocal of the last dilution resulting in at least 50% inhibition.
Time Frame: Prior to, 1 month, 1 year, 2 years, 3 years and 4 years after vaccination.
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 281 | 98
Titer
  Prior to vaccination (N= 255; 83) | 6.3 [5.5 to 7.3] | 5.5 [4.3 to 7.2]
  1 month after vaccination (N= 281; 98) | 482.8 [420.7 to 554.2] | 621.0 [480.3 to 802.9]
  1 year after vaccination (N= 249; 89) | 91.7 [75.6 to 111.3] | 63.8 [43.3 to 94.1]
  2 years after vaccination (N= 235; 86) | 39.3 [31.3 to 49.3] | 30.6 [20.1 to 46.7]
  3 years after vaccination (N= 226; 77) | 29.8 [23.6 to 37.6] | 21.8 [14.2 to 33.5]
  4 years after vaccination (N=208;73) | 5.3 [4.7 to 6.0] | 6.0 [4.5 to 8.0]

6. Secondary Outcome: Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers
Description: Titers are given as Geometric Mean Titers (GMTs). Functional anti-meningococcal serogroup C activity (SBA-MenC) was determined by a serum bactericidal test using rabbit complement. For SBA testing at the PHE at Year 5, titres were expressed as the reciprocal of the last dilution resulting in at least 50% inhibition.
Time Frame: 5 years after vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 195 | 68
Titer | 6.6 [5.6 to 7.8] | 8.5 [5.9 to 12.3]

7. Secondary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Above Cut-off Values
Description: Anti-PRP antibody concentration cut-off values assessed include 0.15 µg/mL (indicative of short-term protection) and 1.0 µg/mL (indicative of long-term protection).
Time Frame: Prior to, 1 month, 1 year, 2 years, 3 years and 4 years after vaccination
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 292 | 100
Subjects
  ≥ 0.15 µg/mL [Prior to vaccination] (N=285,98) | 219 | 82
  ≥ 0.15 µg/mL [1 year post-vaccination] (N=255,91) | 252 | 91
  ≥ 0.15 µg/mL [2 years post-vaccination] (N=237,84) | 235 | 84
  ≥ 0.15 µg/mL [3 years post-vaccination] (N=233,78) | 231 | 77
  ≥ 0.15 µg/mL [4 years post-vaccination] (N=204,73) | 202 | 73
  ≥ 1.0 µg/mL [Prior to vaccination] (N=285,98) | 77 | 22
  ≥ 1.0 µg/mL [1 month post-vaccination] (N=292,100) | 286 | 100
  ≥ 1.0 µg/mL [1 year post-vaccination] (N=255,91) | 209 | 80
  ≥ 1.0 µg/mL [2 years post-vaccination] (N=237,84) | 174 | 72
  ≥ 1.0 µg/mL [3 years post-vaccination] (N=233,78) | 164 | 64
  ≥ 1.0 µg/mL [4 years post-vaccination] (N=204,73) | 144 | 57

8. Secondary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Above Cut-off Values
Description: as for outcome 7
Time Frame: 5 years after vaccination
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 191 | 67
Subjects
  ≥ 0.15 µg/mL [5 years post-vaccination] | 191 | 67
  ≥ 1.0 µg/mL [5 years post-vaccination] | 129 | 47

9. Secondary Outcome: Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs).
Time Frame: Prior to, 1 month , 1 year, 2 years, 3 years and 4 years after vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 292 | 100
microgram per milliliter (µg/mL)
  Prior to vaccination (N=285, 98) | 0.438 [0.374 to 0.512] | 0.472 [0.364 to 0.611]
  1 month after vaccination (N=292, 100) | 46.652 [38.929 to 55.907] | 73.976 [57.624 to 94.968]
  1 year after vaccination (N=255, 91) | 3.550 [2.988 to 4.218] | 4.802 [3.708 to 6.218]
  2 years after vaccination (N= 237, 84) | 2.5 [2.1 to 3.0] | 3.3 [2.5 to 4.2]
  3 years after vaccination (N= 233, 78) | 2.234 [1.886 to 2.647] | 2.751 [2.113 to 3.582]
  4 years after vaccination (N= 204, 73) | 2.116 [1.773 to 2.524] | 2.964 [2.215 to 3.966]

10. Secondary Outcome: Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs).
Time Frame: 5 years after vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 191 | 67
microgram per milliliter (µg/mL) | 2.131 [1.752 to 2.592] | 2.537 [1.815 to 3.546]

11. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentration Above the Cut-off Values
Description: Anti-PSC antibody concentration cut-off values assessed include greater than or equal to (≥) 0.30 µg/mL and ≥ 2.0 µg/mL.
Time Frame: Prior to, 1 month, 1 year, 2 years and 3 years after vaccination
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity (prior to and 1 month after vaccination) and the ATP cohort for analysis of persistence for Year 1, 2, 3 (1, 2, 3 years after vaccination), on subjects with available data for at least one tested antigen at the considered time point.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 290 | 100
Subjects
  ≥ 0.3 µg/mL [prior to vaccination] (N=283, 96) | 2 | 1
  ≥ 0.3 µg/mL [1 month post-vaccination] (N=290,100) | 290 | 100
  ≥ 0.3 µg/mL [1 year post-vaccination] (N=250, 91) | 95 | 33
  ≥ 0.3 µg/mL [2 years post-vaccination] (N=233,84) | 47 | 17
  ≥ 0.3 µg/mL [3 years post-vaccination] (N=230,79) | 24 | 8
  ≥ 2.0 µg/mL [prior to vaccination] (N=283, 96) | 0 | 0
  ≥ 2.0 µg/mL [1 month post-vaccination] (N=290,100) | 289 | 96
  ≥ 2.0 µg/mL [1 year post-vaccination] (N=250, 91) | 6 | 0
  ≥ 2.0 µg/mL [2 years post-vaccination] (N=233,84) | 1 | 1
  ≥ 2.0 µg/mL [3 years post-vaccination] (N=230,79) | 1 | 1

12. Secondary Outcome: Anti-polysaccharide C (Anti-PSC) Antibody Concentrations
Description: Concentrations given as Geometric Mean Concentrations (GMCs).
Time Frame: Prior to, 1 month, 1 year, 2 years and 3 years after vaccination
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 290 | 100
micrograms per milliliter (µg/mL)
  Prior to vaccination (N=283, 96) | NA [NA to NA] — Values were below the assay cut-off at this timepoint of 0.3 µg/mL. | NA [NA to NA] — Values were below the assay cut-off at this timepoint of 0.3 µg/mL.
  1 month after vaccination (N=290,100) | 18.69 [17.10 to 20.42] | 7.95 [6.95 to 9.08]
  1 year after vaccination (N=250, 91) | NA [NA to 0.30] — Lower limits of 95% confidence interval not reliable because of deviation from log normal distribution (large number of imputed values) | NA [NA to NA] — Values were below the assay cut-off at this timepoint of 0.3 µg/mL.
  2 years after vaccination (N= 233, 84) | 0.2 [NA to NA] — Lower and Upper limits of 95% confidence interval not reliable because of deviation from log normal distribution (large number of imputed values) | 0.2 [NA to NA] — Lower and Upper limits of 95% confidence interval not reliable because of deviation from log normal distribution (large number of imputed values)
  3 years after vaccination (N= 230, 79) | NA [NA to NA] — Values were below the assay cutoff at this timepoint of 0.3 μg/mL. | NA [NA to NA] — Values were below the assay cutoff at this timepoint of 0.3 μg/mL.

13. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the injection site.
  Solicited general symptoms assessed include drowsiness, fever (≥ 38°C), irritability and loss of appetite.
Time Frame: Within 4 days (Day 0 -Day 3) after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on vaccinated subjects with available data for the vaccination phase.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 324 | 109
Subjects
  Pain | 91 | 42
  Redness | 146 | 64
  Swelling | 78 | 41
  Drowsiness | 102 | 40
  Fever | 76 | 30
  Irritabily | 154 | 69
  Loss of appetite | 102 | 40

14. Secondary Outcome: Number of Subjects Reporting Unsolicited Symptoms
Description: Unsolicited symptom: Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any solicited symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Time Frame: Within 31 days (Day 0 - Day 30) after vaccination
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 324 | 109
Subjects | 217 | 81

15. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study subject.
  For the long-term persistence phase (Years 1 through 5), only those SAEs that are determined by the investigator to have a causal relationship to the vaccination will be described individually.
Time Frame: Throughout the entire study period (up to year 5)
Population: Analysis was performed on vaccinated subjects from the Total Vaccinated Cohort for the Vaccination Phase of the study (up to Month 1) and on the Total Enrolled Cohort up to Year 5, which included all vaccinated subjects in the vaccination phase who came back for the Year 1, Year 2, Year 3 ,Year 4 and/or Year 5 persistence phases of the study.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 324 | 109
Subjects
  Vaccination Phase (N=324, 109) | 4 | 2
  Until year 5 (N=295, 100) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Year 5 for Serious Adverse Events. Within 31 days after vaccination for Other Adverse Events that were not systematically assessed. Within 4 days after vaccination for Other Adverse Events that were systematically assessed.
Description: For long-term persistence (Years 1 to 5), only SAEs that are determined by the investigator as causally related to vaccination will be described individually. No SAEs related to vaccination were reported between the end of the vaccination phase up to Year 5.
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Serious Adverse Events (participants affected / at risk) | 4/324 | 2/109
Other Adverse Events (participants affected / at risk) | 293/324 | 104/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menitorix Group (N=324) | Meningitec + Hiberix Group (N=109)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Breath holding (Psychiatric disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menitorix Group (N=324) | Meningitec + Hiberix Group (N=109)
Upper respiratory tract infection (Infections and infestations) | 54 | 13
Teething (Gastrointestinal disorders) | 40 | 15
Pyrexia (General disorders) | 37 | 13
Rash (Skin and subcutaneous tissue disorders) | 24 | 17
Diarrhea (Gastrointestinal disorders) | 25 | 8
Vomiting (Gastrointestinal disorders) | 22 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 3
Injection site reaction (General disorders) | 7 | 10
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 9 | 9
Irritability (General disorders) | 0 | 9
Pain (General disorders) | 91 | 42
Redness (General disorders) | 146 | 64
Swelling (General disorders) | 78 | 41
Drowsiness (General disorders) | 102 | 40
Fever (above or equal to 38 degrees Celsius) (General disorders) | 76 | 30
Irritability (General disorders) | 154 | 69
Loss of appetite (General disorders) | 102 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.